CLINICAL TRIAL: NCT06937008
Title: Effect of Whole Body Vibration on Balance in Post Menopause Diabetic Women
Brief Title: Effect Whole Body Vibration on Balance in Post Diabetic Menopause Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahd Tarek Helmy el Dears, Department of Physical Therapy for Women's Health Faculty of Physical Therapy Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cairo university Faculty of PT
Record Dates: First submitted 2025-01-06; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2024-11

CONDITIONS: Diabetic Peripheral Neuropathy; Postmenopausal Women
Keywords: balance; quality of life; whole body vibration; diabetes; postmenopausal
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- WBV group (Experimental): consisted of twenty postmenopausal women with diabetic neuropathy who received whole body vibration and balancing exercise (three times per week for 12 weeks).
  Interventions: Other: Whole body vibration; Other: Balance training
- Balance group (Active Comparator): consisted of twenty postmenopausal women with diabetic neuropathy who received the same balancing exercises as for group A (three times per week for 12 weeks).
  Interventions: Other: Balance training

INTERVENTIONS:
Other: Whole body vibration — All women in group (A) received whole body vibration and balance board training, three times per week for three months.
  Parameters: The WBV was performed by using whole body vibration which is a side-alternating vibration device working as a teeterboard with amplitude of 0 to 5.3 mm (medial to distal) and a variable frequency of 5 to 30 Hz. The amplitude was controlled by adjusting the foot position from 1 to 3, with the larger the position, the greater the amplitude. Before the treatment, procedures of using the Galileo 900 were instructed by the research assistant and its safety issues explained.
  Patient's position: The patient was asked to stand on WBV device by Hold hand support for those elderly women. the vibrating platform in a 100 to 110° squat position, the oscillating platform operating at 20Hz in bare feet at the second foot position for 15 minutes a day for 3 days a week for 3 months. All unusual or uncomfortable complaints from subjects during the WBV treatment were docu
  Arms: WBV group
Other: Balance training — Balance training exercises treatment: All women in both group (A, B) received balance training exercises on balance ball, half ball and balance board exercises three times per week for 3 months

SUMMARY:
Postmenopausal diabetic women have significant balance deficits and increased fall risk. Whole-body vibration may improve balance in these population but needs further research. The purpose of the current study was to determine the effect of whole-body vibration on balance in postmenopausal diabetic women.

DETAILED DESCRIPTION:
Background: Menopause is characterized by reduced androgens produced by ovaries, which negatively affect women health including metabolism and quality of life (QoL) and sexual function. Purpose: This study investigates the effect of whole-body vibration on balance and QoL in postmenopausal diabetic women. Methods: Forty postmenopausal women with diabetic neuropathy will participate in this study aged from 50 to 65 years. They will be randomly distributed into two equal groups: Group A (study group): will receive whole body vibration (WBV) and balancing exercise. Group B (control group): will receive the same balancing exercises as group A. The treatment will be performed 3 times per week for 12 weeks. Dynamic balance will be assessed by Biodex Balance System (BBS) that assesses (Overall stability index [OSI], anteroposterior stability index [APSI] and mediolateral stability index [MLSI)], Berg Balance test (BBT) and Time up and go test (TUG). Quality of life will be assessed by menopous specific in Quality of Life questionnaire before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

Patients were examined by a gynaecologist before the study and were selected according to the following criteria:

* Diabetic postmenopausal women who suffered from peripheral neuropathy
* Their ages ranged from 50 to 65 years.
* Body Mass Indices (BMI) ≤ 30kg/m2
* They were medically stable.

Exclusion Criteria:

* Patients were examined by a gynaecologist before the study and were excluded if they had:

  * Inner ear disturbance.
  * Musculoskeletal problems.
  * Active tuberculosis and tumours.
  * Implanted cardiac rhythm devices.
  * Any hormonal replacement therapy or drug treatment that could affect normal metabolism of musculoskeletal system.
  * Habitual exercise or participate in any supervised exercise.
  * Hypo- or hyperparathyroidism, renal, liver, or chronic disease.

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-05-28 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
OSI | pre and after 3 months of intervention
  TThe BBS measures, in degrees, the tilt about each axis during dynamic conditions and calculates a medial-lateral stability index (MLSI), anterior-posterior stability index (APSI), and an overall stability index (OSI). The OSI score is believed to be the best indicator of the overall ability.

CONTACTS AND LOCATIONS:
Locations (1):
- Haven Police and El Bagour specialized Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No